CLINICAL TRIAL: NCT07085104
Title: A Phase 1 Study Evaluating the Safety and Preliminary Efficacy of ALLO-329, a Dual Anti-CD19/Anti-CD70 Allogeneic CAR T Cell Product in Autoimmune Disease
Brief Title: A Study to Investigate the Safety and Preliminary Efficacy of ALLO-329, an Allogeneic CAR T-cell Therapy, in Adults With Autoimmune Disease
Acronym: RESOLUTION
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allogene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-329-101
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus (With and Without Nephritis); Idiopathic Inflammatory Myopathy; Systemic Sclerosis
Keywords: Systemic lupus erythematosus; SLE; Lupus nephritis; LN; Idiopathic inflammatory myopathy; IIM; Myositis; Dermatomyositis; Anti-synthetase syndrome; Systemic sclerosis; Scleroderma; SSc; Autoimmune disease; CAR T; Allogeneic CAR T; CD19; CD70; AlloCAR T™
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myositis; Scleroderma, Systemic; Lupus Nephritis; Dermatomyositis; Scleroderma, Diffuse; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALLO-329, Cyclophosphamide (Experimental): Participants receive ALLO-329 following lymphodepletion regimen comprised of cyclophosphamide.
  Interventions: Genetic: ALLO-329; Drug: Cyclophophamide
- ALLO-329 (Experimental): Participants receive ALLO-329 without a lymphodepletion regimen.
  Interventions: Genetic: ALLO-329

INTERVENTIONS:
Genetic: ALLO-329 — An allogeneic CAR T cell therapy targeting CD19 and CD70
Drug: Cyclophophamide — Chemotherapy for lymphodepletion
  Arms: ALLO-329, Cyclophosphamide

SUMMARY:
This is a first-in-human, single-arm, open-label study evaluating the safety, tolerability, and preliminary efficacy of ALLO-329 in adults with autoimmune diseases: systemic lupus erythematosus (SLE) with and without renal involvement, idiopathic inflammatory myopathy (IIM), and systemic sclerosis (SSc).The purpose of this trial is to evaluate the safety and tolerability of ALLO-329, an allogeneic anti-CD19, anti-CD70 dual chimeric antigen receptor (CAR) T cell therapy, in adults with autoimmune disorders, provide initial evidence of biological activity and clinical response to the treatment and determine the recommended Phase 2 regimen (RP2R).

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 to < 70 years of age.
2. Adequate hematological function and liver, cardiac, and pulmonary function.
3. A highly sensitive urine pregnancy test or serum pregnancy test (for females of childbearing potential) negative at screening. All participants of childbearing potential must be willing to use a highly effective method of contraception for at least 12 months (6 months for males) after LD chemotherapy or ALLO-329 administration, whichever is later.
4. Signed and dated informed consent form.
5. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures.
6. Confirmed active disease (SLE, IIM, or SSc) as defined by the appropriate classification criteria for each respective disease, clinical evidence, and/or laboratory testing.
7. Disease activity as above despite prior treatment with standard of care therapy including at least one immunosuppressive agent for at least 3 months (in addition to hydroxychloroquine [HCQ]).

Exclusion Criteria:

1. Participants with active systemic bacterial, fungal, or viral infection requiring systemic treatment or a clinically significant active, opportunistic, chronic or recurrent infection.
2. Any active malignancy within 3 years prior to enrollment, except for adequately treated localized basal cell or squamous cell skin cancer, carcinoma in situ or low risk prostate cancer (Gleason score ≤ 6).
3. Prior treatment with CD19 or CD70 targeted therapy or any prior engineered cell therapy (e.g., CAR T therapy).
4. Clinically significant or unstable or uncontrolled acute or chronic disease (e.g., hypothyroidism and diabetes) not due to SLE/IIM/SSc.
5. Symptomatic cardiac or vascular disease requiring medical intervention within 6 months prior to screening, hemodynamically symptomatic pericardial effusion, or symptomatic electrocardiogram abnormality requiring medical intervention.
6. Child-Pugh Class B or C cirrhosis.
7. Symptomatic airway disease requiring medical intervention, pleural effusion ≥ Grade 2, or history of pulmonary embolism requiring anticoagulant therapy within 6 months of enrollment.
8. Participants known to be refractory to platelet or red blood cell transfusions or who will refuse indicated transfusion support to manage cell counts following treatment.
9. Any form of primary, inherited immunodeficiency.
10. Unwilling to participate in an extended safety monitoring period.
11. For participants with SLE: Active disease involving CNS within the last 6 months or SLE that is drug-induced. For those with lupus nephritis, history of dialysis within 12 months or expected need for renal replacement therapy within the next 12 months, or National Institutes of Health (NIH) chronicity score of 3+ in any of the following domains: glomerular sclerosis, glomerular fibrous crescents, tubular atrophy, and/or interstitial fibrosis.
12. Participants with IIM: A myositis other than IIM classification, non-reversible, unrelated or weakness not amenable to assessment, or dermatomyositis with presence of anti-TIF1 gamma antibody.
13. Participants with SSc: Pulmonary arterial hypertension requiring treatment, rapidly progressive or severe SSc gastrointestinal involvement, or prior scleroderma renal crisis.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting toxicities (DLTs) and Other Safety Parameters | Up to 60 months
  The incidence of dose limiting toxicities (DLTs) and other safety parameters (including but not limited to treatment emergent adverse events [AEs], serious adverse events [SAEs], and clinical laboratory abnormalities)

SECONDARY OUTCOMES:
Disease Response to Treatment - Systemic Lupus Erythematosus | Up to 60 months
  Efficacy as assessed by rates of achieving SRI-4, LLDAS and DORIS remission.
Disease Response to Treatment - Systemic Lupus Erythematosus | Up to 60 months
  Efficacy as assessed by change from baseline in SLEDAI-2K score.
Disease Response to Treatment - Lupus Nephritis | Up to 60 months
  Efficacy as assessed by complete renal response (CRR) and partial renal response (PRR).
Disease Response to Treatment - Idiopathic Inflammatory Myopathy | Up to 60 months
  Efficacy as assessed by ACR/EULAR myositis response criteria components.
Disease Response to Treatment - Systemic Sclerosis | Up to 60 months
  Efficacy as assessed by change from baseline in the European Scleroderma Trials and Research Group (EUSTAR) activity index.
Disease Response to Treatment - Systemic Sclerosis | Up to 60 months
  Efficacy as assessed by change from baseline in the American College of Rheumatology Composite Response Index in Diffuse Cutaneous Systemic Sclerosis (ACR-CRISS).
ALLO-329 Peak Expansion (Cmax) | Up to 60 months
ALLO-329 Persistence Over Time Including Area Under the Expansion Curve (AUC) | Up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Allogene Study Director, Study Director — Allogene Therapeutics, Inc.
Locations (10):
- United States (9):
  - Mayo Clinic, Phoenix, Arizona
  - University of Iowa, Iowa City, Iowa
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Astera Cancer Care, East Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health, Greenville, South Carolina
  - LDS Hospital - lntermountain Health, Salt Lake City, Utah
- Hôpital Maisonneuve Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No